CLINICAL TRIAL: NCT04875949
Title: Anti-Cholinergic Receptors Antibodies and Dysautonomia Symptoms Relationships in Pure Autonomic Failure, Amyotrophic Lateral Sclerosis, Postural Orthostatic Tachycardia Syndrome: a Pathophysiology Based Therapeutic New Strategy.
Brief Title: Anti-Cholinergic Receptors Antibodies, Autonomic Profile and Dysautonomia Symptoms in PAF, ALS and POTS (DISAUT-AB)
Acronym: DISAUT-AB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Fondazione Salvatore Maugeri (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DISAUT-AB ICH
Record Dates: First submitted 2021-01-12; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pure Autonomic Failure; Amyotrophic Lateral Sclerosis; Postural Orthostatic Tachycardia Syndrome; Anti-Cholinergic Receptors Antibodies
Keywords: Neural control of circulation and respiration; Anti-Cholinergic receptors antibodies; Power Spectrum Analysis
MeSH Terms: conditions — Pure Autonomic Failure; Amyotrophic Lateral Sclerosis; Postural Orthostatic Tachycardia Syndrome; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-AChRs Abs positive patients (Experimental): Immunoabsorption
  Interventions: Procedure: Immunoabsorption/plasmapheresis procedure

INTERVENTIONS:
Procedure: Immunoabsorption/plasmapheresis procedure

SUMMARY:
Anti alfa-3 and alfa-7 ganglionic cholinergic receptors (anti-AChRs) antibodies (Abs) plasma removal by plasmapheresis (1,2) acutely improved dysautonomia symptoms in case reports with Pure Autonomic Failure (PAF) (3). We shall assess the prevalence of anti-AChRs Ab and the relationship among Ab titer, cardiovascular autonomic profile and symptoms in neurodegenerative diseases characterized by similar dysautonomia symptoms such as PAF, Amyotrophic Lateral Sclerosis (ALS) and Postural Orthostatic Tachycardia Syndrome (POTS) (4). Ab positive patients will undergo selective immunoabsorption once a week up to achievement of Ab titer lower than 65% of baseline followed by immunosuppressive therapy with prednisone. Both Ab positive and negative groups will undergo anti-AChR Abs, autonomic profile and dysautonomia symptoms assessment, every 4 months up to 3 years. Evidence of correlation among reduced Ab titer and autonomic profile and symptoms improvement may result in new effective therapy.

DETAILED DESCRIPTION:
PAF is a rare neurodegenerative disorder characterized by symptoms due to sympathetic failure, such as orthostatic hypotension and syncope, and deficient parasympathetic activity such as constipation, urinary retention and decreased salivation (3). Plasma anti-AChRs Abs were found in PAF (1, 2, 5) and in POTS (6), raising the possibility that Ab mediated alterations in the ganglionic cholinergic function might induce autonomic abnormalities and related symptoms. Anti-AchRs Abs removal by plasmapheresis was associated with acute improvement of orthostatic tolerance in PAF single case report (2).

There is no data on the medium/long term clinical follow-up of these patients. Nothing is known about the time course of the relationships among Abs plasma titer, neural autonomic profile and symptoms if a selective immunoabsorption procedure is combined with drug immunosoppression (Prednisone) to lower Ab levels and potentially ameliorate ganglionic function.

Finally, it is unknown whether a neurodegenerative disease with concomitant dysautonomia symptoms such as the Amyotrophic Lateral Sclerosis (ALS) may share an analogous anti-AChRs Ab profile. Variations in cholinergic receptor subunits 3 and 4 were observed in ALS but no plasma anti-AChRs Abs were searched for (7). Abs removal by immunoabsorption technique combined with drug immunosoppression might represent a new effective therapy for dysautonomia symptoms in ALS as well as in POTS and PAF.

Hyphotesis and Significance:

* Changes in anti-AChR Abs plasma titer may be mirrored by modifications in the cardiovascular autonomic profile, as assessed by spectrum analysis of RR and arterial pressure variability, and be related to fluctuations in the magnitude of dysautonomia symptoms in PAF, ALS and POTS patients.
* Plasma anti-AChR Abs might underlie dysautonomia symptoms associated to neurodegenerative disorders such as ASL and POTS
* Plasma anti-AChR Abs removal by selective immunoabsorption techniques may improve ganglionic transmission leading to clinical amelioration and represent a new effective etiologic therapy for these diseases.

Specific Aim:

Aim 1: To evaluate the prevalence of plasma anti-AChR Abs in patients affected by PAF, ALS and POTS .

Aim 2: To address the time course and relationships of anti-AChR Abs plasma titers, cardiovascular autonomic profile and dysautonomia symptoms before and after anti-AChR Abs plasma removal by selective immunoabsorption technique in PAF, ALS and POTS patients. The core laboratory of the Neuroimmunology Unit of Istituto Neurologico Besta will provide expertise and facilities for assessing plasma anti-AChR Abs. The clinical laboratory of Clinica Medica Syncope Unit (Humanitas) will provide the know-how and facilities for patients neural autonomic assessment.

Aim 3:To set up a new therapeutic strategy based on selective immunoabsorption technique sessions combined with drug immunosuppression (Prednisone) in patients with anti-AChR Abs.

ELIGIBILITY:
Inclusion Criteria:

• Patients, older than 18 years affected by PAF, ALS and POTS, with dysautonomia symptoms assessed by clinical evaluation and by the Composite Autonomic Scoring Scale (CASS)

Exclusion Criteria:

* Hepatic, renal, heart and other secondary causes of autonomic dysfunction
* History/familiarity with seizures
* Atrial fibrillation and other relevant cardiac rhythm disturbances
* Diabetes
* Other neurological or psychiatric diseases
* Pacemakers or other electronic implants inserted into the body
* Coronary disorders, elevated intracranial blood pressure
* Assumption of drugs facilitating seizures, psychiatric drugs, alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of plasma anti-AChR Abs in PAF, ALS and POTS | 3 years
  Number of patients with plasma anti-AChR Abs
Effects of anti-AChR Abs removal on dysautonomic symptoms | 3 years
  COMPASS31 scores (range 0-100; 0 best -100 worst)
Time course of dysautonomia symptoms | 3 years
  COMPASS31 scores (range: 0-100; 0 best-100 worst)
Time course of orthostatic tolerance | 3 years
  Orthostatic tolerance (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaello Furlan, Prof., Principal Investigator — Humanitas Research Hospital, Humanitas University; Franca Barbic, MD, Study Chair — Humanitas Research Hospital, Humanitas University, Rozzano; Raffaello Furlan, Prof., Study Director — Humanitas Research Hospital, Humanitas University
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy

REFERENCES:
- [Background] Vernino S, Low PA, Fealey RD, Stewart JD, Farrugia G, Lennon VA. Autoantibodies to ganglionic acetylcholine receptors in autoimmune autonomic neuropathies. N Engl J Med. 2000 Sep 21;343(12):847-55. doi: 10.1056/NEJM200009213431204. PMID 10995864
- [Background] Schroeder C, Vernino S, Birkenfeld AL, Tank J, Heusser K, Lipp A, Benter T, Lindschau C, Kettritz R, Luft FC, Jordan J. Plasma exchange for primary autoimmune autonomic failure. N Engl J Med. 2005 Oct 13;353(15):1585-90. doi: 10.1056/NEJMoa051719. PMID 16221781
- [Background] Furlan R, Jacob G, Snell M, Robertson D, Porta A, Harris P, Mosqueda-Garcia R. Chronic orthostatic intolerance: a disorder with discordant cardiac and vascular sympathetic control. Circulation. 1998 Nov 17;98(20):2154-9. doi: 10.1161/01.cir.98.20.2154. PMID 9815870
- [Background] Vernino S, Hopkins S, Wang Z. Autonomic ganglia, acetylcholine receptor antibodies, and autoimmune ganglionopathy. Auton Neurosci. 2009 Mar 12;146(1-2):3-7. doi: 10.1016/j.autneu.2008.09.005. Epub 2008 Oct 31. PMID 18951069
- [Background] Sabatelli M, Eusebi F, Al-Chalabi A, Conte A, Madia F, Luigetti M, Mancuso I, Limatola C, Trettel F, Sobrero F, Di Angelantonio S, Grassi F, Di Castro A, Moriconi C, Fucile S, Lattante S, Marangi G, Murdolo M, Orteschi D, Del Grande A, Tonali P, Neri G, Zollino M. Rare missense variants of neuronal nicotinic acetylcholine receptor altering receptor function are associated with sporadic amyotrophic lateral sclerosis. Hum Mol Genet. 2009 Oct 15;18(20):3997-4006. doi: 10.1093/hmg/ddp339. Epub 2009 Jul 23. PMID 19628475
- [Background] Vernino S, Adamski J, Kryzer TJ, Fealey RD, Lennon VA. Neuronal nicotinic ACh receptor antibody in subacute autonomic neuropathy and cancer-related syndromes. Neurology. 1998 Jun;50(6):1806-13. doi: 10.1212/wnl.50.6.1806. PMID 9633732
- [Background] Furlan R, Piazza S, Bevilacqua M, Turiel M, Norbiato G, Lombardi F, Malliani A. Pure Autonomic Failure: complex abnormalities in the neural mechanisms regulating the cardiovascular system. J Auton Nerv Syst. 1995 Mar 2;51(3):223-35. doi: 10.1016/0165-1838(94)00135-7. PMID 7769156
- [Background] Barbic F, Perego F, Canesi M, Gianni M, Biagiotti S, Costantino G, Pezzoli G, Porta A, Malliani A, Furlan R. Early abnormalities of vascular and cardiac autonomic control in Parkinson's disease without orthostatic hypotension. Hypertension. 2007 Jan;49(1):120-6. doi: 10.1161/01.HYP.0000250939.71343.7c. Epub 2006 Nov 13. PMID 17101845
- [Background] Porta A, Castiglioni P, Di Rienzo M, Bari V, Bassani T, Marchi A, Takahashi AC, Tobaldini E, Montano N, Catai AM, Barbic F, Furlan R, Cividjian A, Quintin L. Short-term complexity indexes of heart period and systolic arterial pressure variabilities provide complementary information. J Appl Physiol (1985). 2012 Dec 15;113(12):1810-20. doi: 10.1152/japplphysiol.00755.2012. Epub 2012 Oct 25. PMID 23104699
- [Background] Furlan R, Porta A, Costa F, Tank J, Baker L, Schiavi R, Robertson D, Malliani A, Mosqueda-Garcia R. Oscillatory patterns in sympathetic neural discharge and cardiovascular variables during orthostatic stimulus. Circulation. 2000 Feb 29;101(8):886-92. doi: 10.1161/01.cir.101.8.886. PMID 10694528
- [Background] Barbic F, Galli M, Dalla Vecchia L, Canesi M, Cimolin V, Porta A, Bari V, Cerri G, Dipaola F, Bassani T, Cozzolino D, Pezzoli G, Furlan R. Effects of mechanical stimulation of the feet on gait and cardiovascular autonomic control in Parkinson's disease. J Appl Physiol (1985). 2014 Mar 1;116(5):495-503. doi: 10.1152/japplphysiol.01160.2013. Epub 2014 Jan 16. PMID 24436294
- [Background] Low PA. Composite autonomic scoring scale for laboratory quantification of generalized autonomic failure. Mayo Clin Proc. 1993 Aug;68(8):748-52. doi: 10.1016/s0025-6196(12)60631-4. PMID 8392653
- [Background] Chio A, Mora G, Restagno G, Brunetti M, Ossola I, Barberis M, Ferrucci L, Canosa A, Manera U, Moglia C, Fuda G, Traynor BJ, Calvo A. UNC13A influences survival in Italian amyotrophic lateral sclerosis patients: a population-based study. Neurobiol Aging. 2013 Jan;34(1):357.e1-5. doi: 10.1016/j.neurobiolaging.2012.07.016. Epub 2012 Aug 22. PMID 22921269
- [Background] Chio A, Calvo A, Moglia C, Mazzini L, Mora G; PARALS study group. Phenotypic heterogeneity of amyotrophic lateral sclerosis: a population based study. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):740-6. doi: 10.1136/jnnp.2010.235952. Epub 2011 Mar 14. PMID 21402743